CLINICAL TRIAL: NCT03325712
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 705564 (Double-blind, Randomised, Placebo-controlled, Parallel-group Design) and Evaluation of Midazolam Interaction (Nested, Open, Fixed-sequence, Intra-individual Comparison) in Healthy Male Subjects
Brief Title: This Study in Healthy Men Tests How Different Doses of BI 705564 Are Taken up in the Body and How Well They Are Tolerated. The Study Also Tests How BI 705564 Affects the Way the Body Breaks Down Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1408-0002; 2017-003269-85 (EudraCT Number)
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Results first posted 2022-07-11 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-07

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Dose group 1: BI 705564 10 mg (Experimental)
  Interventions: Drug: BI 705564
- Dose group 2: BI 705564 20 mg (Experimental)
  Interventions: Drug: BI 705564; Drug: Midazolam
- Dose group 3: BI 705564 40 mg (Experimental)
  Interventions: Drug: BI 705564; Drug: Midazolam
- Dose group 5: BI 705564 60 mg (Experimental)
  Interventions: Drug: BI 705564; Drug: Midazolam
- Dose group 4: BI 705564 80 mg (Experimental)
  Interventions: Drug: BI 705564; Drug: Midazolam
- Placebo matching BI 705564 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Midazolam
- Dose group 8: BI 705564 40 mg - SPT (Experimental): SPT stands for skin prick test.
  Interventions: Drug: BI 705564
- Placebo matching BI 705564 - SPT (Placebo Comparator): SPT stands for skin prick test.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 705564 — Film-coated tablet
  Arms: Dose group 1: BI 705564 10 mg; Dose group 2: BI 705564 20 mg; Dose group 3: BI 705564 40 mg; Dose group 4: BI 705564 80 mg; Dose group 5: BI 705564 60 mg; Dose group 8: BI 705564 40 mg - SPT
Drug: Placebo — Film-coated tablet
  Arms: Placebo matching BI 705564; Placebo matching BI 705564 - SPT
Drug: Midazolam — Solution for injection
  Arms: Dose group 2: BI 705564 20 mg; Dose group 3: BI 705564 40 mg; Dose group 4: BI 705564 80 mg; Dose group 5: BI 705564 60 mg; Placebo matching BI 705564

SUMMARY:
The primary objective of this trial is to investigate safety and tolerability of BI 705564 in healthy male subjects, following oral administration of multiple rising doses.

Secondary objectives are the exploration of the pharmacokinetics, including dose proportionality and investigation of linearity.

ELIGIBILITY:
Inclusion Criteria:

* Dose Groups (DGs)1 to 5: Healthy male subjects according to the assessment of the investigator, based on a complete medical history, a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests;
* DG 8, only: Otherwise healthy male subjects (as defined for DGs 1 to 5) with a history (of at least 1 year) of IgE-mediated, perennial allergies, predominantly to (house) dust mite (dermatophagoides pteronyssinus or dermatophagoides farina) as documented by a positive Skin prick test (SPT)(largest diameter of wheal at screening > 5 mm)

  * Age of 18 to 50 years (incl.)
  * Body Max Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
  * Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/ or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizure or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication, if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug.
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to the administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

* Male subject with women of child bearing potential (WOCBP) partner who is unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication
* Subjects who, in the investigator's judgement, are perceived as having an increased risk of bleeding, e.g. history of haemorrhagic disorders, clinical relevant petechial bleeding, occult blood in faeces, haematuria in repeated urine tests, trauma or surgery within the last month planned surgery during trial participation, history of arteriovenous malformation or aneurysm, history of gastroduodenal ulcer disease or gastrointestinal haemorrhage, history of intracranial, intraocular, spinal, retroperitoneal, or atraumatic intraarticular bleeding, use of drugs that may interfere with haemostasis during trial conduct (e.g. acetylic salicylic acid or other non-steroidal anti-inflammatory drugs)
* Repeated platelet counts below 100 cells/nL at screening
* Bleeding times (to monitor platelet function) above reference range at screening
* Repeated absolute B cell (CD19+) counts below 40/μL at screening
* Serum potassium below normal range at screening
* A history or current clinical signs of acute pancreatitis
* Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The evaluation of multiple rising dose (MRD) of BI 705564 was designed as randomised, placebo-controlled, double-blind and parallel-group design and the evaluation of midazolam interaction was designed as nested, open-label, fixed-sequence, intra-individual comparison in healthy male participants.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist sites which would then ensured that all participants met all strictly inclusion/exclusion criteria. Participants were not to be assigned to treatment groups if any of the specific entry criteria were violated.
Groups:
- Placebo Matching BI 705564: Participants were orally administered placebo matching to BI 705564 film-coated tablets (and 75 microgram (μg) Midazolam solution for injection, for dose groups 2-5) with 240 milliliter (mL) of water after a standard continental breakfast, on Day 1 and once per day on Days 4 to 17 (for placebo) and on Day -1 and Day 17 (for Midazolam).
- Placebo Matching BI 705564 - SPT: Participants with a positive skin prick test (SPT) were orally administered once daily for 28 days placebo matching to BI 705564 film-coated tablets with 240 milliliter (mL) of water after breakfast.
- Dose Group 1: BI 705564 10 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 1 film-coated tablet of 10 milligram (mg) of BI 705564 with 240 milliliter (mL) of water after a standard continental breakfast.
- Dose Group 2: BI 705564 20 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 2 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=20 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (μg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
- Dose Group 3: BI 705564 40 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 4 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=40 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (μg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
- Dose Group 5: BI 705564 60 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 6 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=60 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (μg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
- Dose Group 4: BI 705564 80 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 8 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=80 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (µg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
- Dose Group 8: BI 705564 40 mg - SPT: Participants with a positive skin prick test (SPT) were orally administered for 28 days once daily 4 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=40 mg) with 240 milliliter (mL) of water after breakfast.
Period: Overall Study
Arm/Group | Placebo Matching BI 705564 | Placebo Matching BI 705564 - SPT | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
Started | 10 | 2 | 8 | 8 | 8 | 8 | 8 | 8
Completed | 10 | 2 | 8 | 8 | 6 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): This subject set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 705564 | Placebo Matching BI 705564 - SPT | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT | Total
Number analyzed (Participants) | 10 | 2 | 8 | 8 | 8 | 8 | 8 | 8 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (8.2) | 33.0 (2.8) | 34.8 (9.6) | 44.0 (5.7) | 32.3 (9.1) | 38.4 (8.3) | 40.5 (10.2) | 28.5 (10.7) | 36.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 2 | 8 | 8 | 8 | 8 | 8 | 8 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 2 | 8 | 8 | 8 | 8 | 8 | 8 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  White | 10 | 1 | 7 | 8 | 8 | 7 | 7 | 7 | 55
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events
Description: Percentage of participants with drug-related adverse events is reported.
Time Frame: From first drug administration until 10 days after last drug administration, up to 27 days (for dose groups 1 to 5 and "Placebo Matching BI 705564") or up to 37 days (for dose group 8 and "Placebo Matching BI 705564 - SPT").
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants (%)
Groups:
- Dose Group 4: BI 705564 80 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 8 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=80 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (μg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
Arm/Group | Placebo Matching BI 705564 | Placebo Matching BI 705564 - SPT | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
Number analyzed (Participants) | 10 | 2 | 8 | 8 | 8 | 8 | 8 | 8
Percentage of participants (%) | 20.0 | 50.0 | 12.5 | 0.0 | 50.0 | 50.0 | 12.5 | 75.0

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 705564 in Plasma Over a Uniform Dosing Interval τ After Administration of the First Dose (AUCτ,1)
Description: Area under the concentration-time curve of BI 705564 in plasma over a uniform dosing interval τ after administration of the first dose of BI 705564 (AUCτ,1) is reported. Here AUCτ,1 = AUC0-24.
Time Frame: 1 hour(s) (h) prior drug administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h after first BI 705564 dose (for dose groups 1 to 5); 1.5 h prior drug administration and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 23 h after first BI 705564 dose (for dose group 8).
Population: Pharmacokinetic (PK) parameter analysis set (PKS) included all subjects in the TS who provided at least one PK parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/liter (nmol*h/L)
Arm/Group | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
nanomole*hour/liter (nmol*h/L) | 42.1 (40.6) | 70.8 (31.7) | 131.0 (22.4) | 168.0 (40.1) | 238.0 (46.6) | 120.0 (33.9)
Statistical Analysis 1: Comparison: Dose Group 1: BI 705564 10 mg vs Dose Group 2: BI 705564 20 mg vs Dose Group 3: BI 705564 40 mg vs Dose Group 5: BI 705564 60 mg vs Dose Group 4: BI 705564 80 mg; The basic model for the investigation of dose proportionality is a power model that describes the functional relationship between the dose and PK endpoints. Statistical hypotheses were not tested in a confirmatory sense; Test type: Other; Slope = 0.8188, 90% CI 2-sided [0.6966 to 0.9410], Standard Error of Mean 0.0725 — Based on the estimate for slope parameter (β), a 2-sided 90% CI for the slope was computed. Perfect dose proportionality would correspond to a slope of 1. Standard error of mean is standard error of slope

3. Secondary Outcome: Maximum Measured Concentration of BI 705564 in Plasma (Cmax) After the Administration of the First Dose
Description: Maximum measured concentration of BI 705564 in plasma (Cmax) after the administration of the first dose of BI 705564 is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Groups:
- Dose Group 2: BI 705564 20 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 2 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=20 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (µg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
- Dose Group 3: BI 705564 40 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 4 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=40 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (µg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
- Dose Group 5: BI 705564 60 mg: Participants were orally administered one single dose on Day 1 and once daily on Days 4 to 17, 6 film-coated tablets of 10 milligram (mg) of BI 705564 (total dosage=60 mg) with 240 milliliter (mL) of water after a standard continental breakfast. On Day -1 and on Day 17 participants were orally administered also 75 microgram (µg) of solution for injection of midazolam with 240 mL of water after a standard continental breakfast.
Arm/Group | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
nanomole/Liter (nmol/L) | 11.4 (42.2) | 18.8 (38.2) | 36.5 (17.8) | 41.0 (28.1) | 58.1 (54.4) | 31.7 (35.2)
Statistical Analysis 1: Comparison: Dose Group 1: BI 705564 10 mg vs Dose Group 2: BI 705564 20 mg vs Dose Group 3: BI 705564 40 mg vs Dose Group 5: BI 705564 60 mg vs Dose Group 4: BI 705564 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.7708, 90% CI 2-sided [0.6449 to 0.8967], Standard Error of Mean 0.0747 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 705564 in Plasma at Steady State Over a Uniform Dosing Interval τ (AUCτ,ss) After the Administration of the Last Dose
Description: Area under the concentration-time curve of BI 705564 in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) after the administration of the last dose of BI 705564 is reported.
  As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: 1 h before last dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h after last BI 705564 dose on Day 17 (for dose groups 1 to 5); 1.5 h before last dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 23 h after last BI 705564 dose on Day 28 (for dose group 8).
Population: Pharmacokinetic (PK) parameter analysis set (PKS) included all subjects in the TS who provided at least one PK parameter that was not excluded. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole *hour/liter (nmol*h/L)
Arm/Group | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
Number analyzed (Participants) | 8 | 8 | 6 | 8 | 8 | 8
nanomole *hour/liter (nmol*h/L) | 45.9 (34.2) | 84.8 (25.9) | 164.0 (34.3) | 170.0 (62.1) | 204.0 (179.0) | 138.0 (32.1)
Statistical Analysis 1: Comparison: Dose Group 1: BI 705564 10 mg vs Dose Group 2: BI 705564 20 mg vs Dose Group 3: BI 705564 40 mg vs Dose Group 5: BI 705564 60 mg vs Dose Group 4: BI 705564 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.7167, 90% CI 2-sided [0.4922 to 0.9412], Standard Error of Mean 0.1330 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Maximum Measured Concentration of BI 705564 in Plasma at Steady State Over a Uniform Dosing Interval τ (Cmax,ss) After the Administration of the Last Dose
Description: Maximum measured concentration of BI 705564 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) after the administration of the last dose.
  As per the protocol, day is counted as "Day 1 = 0:00".
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
Number analyzed (Participants) | 8 | 8 | 6 | 8 | 8 | 8
nanomole/Liter (nmol/L) | 13.3 (29.4) | 19.8 (23.7) | 41.8 (21.4) | 43.4 (57.2) | 52.6 (201.0) | 39.2 (28.3)
Statistical Analysis 1: Comparison: Dose Group 1: BI 705564 10 mg vs Dose Group 2: BI 705564 20 mg vs Dose Group 3: BI 705564 40 mg vs Dose Group 5: BI 705564 60 mg vs Dose Group 4: BI 705564 80 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; Slope = 0.6825, 90% CI 2-sided [0.4556 to 0.9094], Standard Error of Mean 0.1344 — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Area Under the Concentration-time Curve of Midazolam in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) After the First and Last Dose
Description: Area under the concentration-time curve of Midazolam in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) after the first and last dose for "Placebo Matching BI 705564" group and for dose groups 2 to 5 is reported.
Time Frame: 1.5 h prior midazolam administration and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6 and 8 h after first midazolam dose on Day -1 and 1h prior midazolam administration and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6 and 8 h after last midazolam dose on Day 17.
Population: Pharmacokinetic (PK) parameter analysis set (PKS)-midazolam set (PKS-Mida): This set included all subjects in dose groups 2 to 5 who received midazolam (including placebo-treated subjects). Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Least Squares Mean (Standard Error); unit: picomole*hour/Liter (pmol*h/L)
Arm/Group | Placebo Matching BI 705564 | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
picomole*hour/Liter (pmol*h/L)
  After last dose: Midazolam + BI705564 or Midazolam + Placebo (Treatment (T)): number analyzed (Participants) | 8 | 8 | 6 | 8 | 8
  After last dose: Midazolam + BI705564 or Midazolam + Placebo (Treatment (T)) | 4478.58 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.10 | 3463.24 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.06 | 4812.45 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.11 | 3458.32 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.29 | 3759.20 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.10
  After first dose: Midazolam alone (Reference (R)) | 4356.03 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.10 | 3721.70 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.06 | 4382.24 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.1 | 3191.16 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.29 | 3445.42 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.10
Statistical Analysis 1: Comparison: Placebo Matching BI 705564; Placebo matching BI 705564. Relative bioavailability of midazolam is analyzed using analysis of variance (ANOVA) model on logarithmic scale including random effects for "subjects" and fixed effects for "time point"; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 102.81, 90% CI 2-sided [87.18 to 121.25], Standard Deviation 17.5 — The effect of BI 705564 on midazolam is estimated by the ratio of the geometric mean (T/R) and confidence interval (CI). CI is calculated based on the residual error from ANOVA
Statistical Analysis 2: Comparison: Dose Group 2: BI 705564 20 mg; BI 705564 dose group 2. Relative bioavailability of midazolam is analyzed using analysis of variance (ANOVA) model on logarithmic scale including random effects for "subjects" and fixed effects for "time point"; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 93.06, 90% CI 2-sided [79.94 to 108.32], Standard Deviation 17.4 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Dose Group 3: BI 705564 40 mg; BI 705564 dose group 3. Relative bioavailability of midazolam is analyzed using analysis of variance (ANOVA) model on logarithmic scale including random effects for "subjects" and fixed effects for "time point"; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 109.82, 90% CI 2-sided [103.59 to 116.42], Standard Deviation 5.0 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Dose Group 5: BI 705564 60 mg; BI 705564 dose group 5. Relative bioavailability of midazolam is analyzed using analysis of variance (ANOVA) model on logarithmic scale including random effects for "subjects" and fixed effects for "time point"; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio ( T/R) = 108.37, 90% CI 2-sided [92.00 to 127.66], Standard Deviation 17.4 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Dose Group 4: BI 705564 80 mg; BI 705564 dose group 4. Relative bioavailability of midazolam is analyzed using analysis of variance (ANOVA) model on logarithmic scale including random effects for "subjects" and fixed effects for "time point"; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 109.11, 90% CI 2-sided [92.43 to 128.79], Standard Deviation 17.6 — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Maximum Measured Concentration of Midazolam in Plasma (Cmax) After the First and Last Dose
Description: Maximum measured concentration of Midazolam in plasma (Cmax) after the first and last dose for "Placebo Matching BI 705564" group and for dose groups 2 to 5 is reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Least Squares Mean (Standard Error); unit: picomole/Liter (pmol/L)
Arm/Group | Placebo Matching BI 705564 | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
picomole/Liter (pmol/L)
  After last dose: Midazolam +BI 705564 or Midazolam +Placebo (Treatment (T)): number analyzed (Participants) | 8 | 8 | 6 | 8 | 8
  After last dose: Midazolam +BI 705564 or Midazolam +Placebo (Treatment (T)) | 1197.89 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.10 | 1040.42 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.09 | 1255.36 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.11 | 984.14 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.26 | 1058.32 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.11
  After first dose: Midazolam alone (Reference (R)) | 1196.63 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.10 | 1232.26 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.09 | 1147.40 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.11 | 1031.18 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.26 | 1175.41 (NA) — Standard error is actually adjusted geometric standard error. Geometric standard error=1.11
Statistical Analysis 1: Comparison: Placebo Matching BI 705564; [analysis description as in outcome 6, analysis 1]; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 100.10, 90% CI 2-sided [83.99 to 119.31], Standard Deviation 18.7 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Dose Group 2: BI 705564 20 mg; [analysis description as in outcome 6, analysis 2]; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 84.43, 90% CI 2-sided [72.29 to 98.62], Standard Deviation 16.5 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Dose Group 3: BI 705564 40 mg; [analysis description as in outcome 6, analysis 3]; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 109.41, 90% CI 2-sided [94.34 to 126.88], Standard Deviation 13.1 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Dose Group 5: BI 705564 60 mg; [analysis description as in outcome 6, analysis 4]; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 95.44, 90% CI 2-sided [79.75 to 114.21], Standard Deviation 19.1 — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Dose Group 4: BI 705564 80 mg; [analysis description as in outcome 6, analysis 5]; Test type: Other; Standard deviation is intra-individual geometric coefficient of variation (%); Ratio (T/R) = 90.04, 90% CI 2-sided [70.75 to 114.59], Standard Deviation 25.9 — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 10 days after last drug administration, up to 27 days (for dose groups 1 to 5 and "Placebo Matching BI 705564" ) or up to 37 days (for dose group 8 and "Placebo Matching BI 705564 - SPT").
Description: Treated Set (TS): This subject set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Placebo Matching BI 705564 | Placebo Matching BI 705564 - SPT | Dose Group 1: BI 705564 10 mg | Dose Group 2: BI 705564 20 mg | Dose Group 3: BI 705564 40 mg | Dose Group 5: BI 705564 60 mg | Dose Group 4: BI 705564 80 mg | Dose Group 8: BI 705564 40 mg - SPT
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/10 | 2/2 | 3/8 | 2/8 | 4/8 | 5/8 | 2/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 705564 (N=10) | Placebo Matching BI 705564 - SPT (N=2) | Dose Group 1: BI 705564 10 mg (N=8) | Dose Group 2: BI 705564 20 mg (N=8) | Dose Group 3: BI 705564 40 mg (N=8) | Dose Group 5: BI 705564 60 mg (N=8) | Dose Group 4: BI 705564 80 mg (N=8) | Dose Group 8: BI 705564 40 mg - SPT (N=8)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT03325712/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03325712/SAP_001.pdf